CLINICAL TRIAL: NCT02302794
Title: Prospective Randomized Controlled Multicenter Clinical Trial for Comparison of Long-term Outcomes Between Laparoscopy-assisted and Open Distal Subtotal Gastrectomy With D2 Lymphadenectomy for Locally Advanced Gastric Cancer
Brief Title: A Multicenter Clinical Trial on Laparoscopic Gastric Cancer Surgery Compared With Open Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cai Kailin (Other)
Responsible Party: Sponsor-Investigator, Cai Kailin, Associate chief physician of gastrointestinal surgery, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR-TRC-14004877
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2014-11-27 (Estimated); Status verified 2014-07

CONDITIONS: Locally Advanced Gastric Cancer
MeSH Terms: interventions — Conversion to Open Surgery; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- open surgery (Active Comparator): Conventional procedure
  Interventions: Procedure: open surgery
- laparoscopic surgery (Experimental): Minimum invasive procedure
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: open surgery — Patients in this arm undergo radical resection of gastric cancer in open surgery.Open surgery is a conventional technique for gastric cancer patients.
  Other Names: group A; open
  Arms: open surgery
Procedure: laparoscopic surgery — Patients in this arm undergo radical resection of gastric cancer in laparoscopic surgery.Laparoscopic surgery is a new and minimum invasive technique for gastric cancer patients.
  Other Names: group B; laparoscopic
  Arms: laparoscopic surgery

SUMMARY:
evaluate the long-term efficacy and safety of oncology between D2 laparoscopic approach distal gastric resection (distal gastrectomy, D2 lymph node dissection) with the current standard surgical treatment model D2 open approach distal gastric resection (distal gastrectomy, D2 lymphadenectomy).

DETAILED DESCRIPTION:
Study type：Interventional Study phase：Phase III Objectives of Study：to evaluate the long-term efficacy and safety of oncology between D2 laparoscopic approach distal gastric resection (distal gastrectomy, D2 lymph node dissection) with the current standard surgical treatment model D2 open approach distal gastric resection (distal gastrectomy, D2 lymphadenectomy).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years ~ 75 years;
2. the primary adenocarcinoma (papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, signet ring cell carcinoma, poorly differentiated adenocarcinoma);
3. clinical stage T2-4a, N0-3, M0 (according to AJCC-7th TNM staging);
4. to perform distal gastrectomy, D2 lymph node dissection surgical can obtain R0 resection (multiple primary cancers also apply)
5. ECOG performance status 0/1;
6. ASA score I-III;
7. patient informed consent.

Exclusion Criteria:

1. pregnant or lactating women;
2. serious mental illness;
3. upper abdominal surgery (except laparoscopic cholecystectomy );
4. gastric surgery (including for gastric ESD / EMR);
5. imaging examinations showed regional integration lymph nodes (maximum diameter ≥ 3cm)
6. other malignant diseases in 5 years;
7. implemented or recommended neoadjuvant therapy in patients with gastric cancer ;
8. have unstable angina or myocardial infarction within six months; (9) have cerebral infarction or cerebral hemorrhage within 6 months; (10) sustained systemic glucocorticoid treatment history within 1 month; (11) have other diseases needed operative treatment at the same time; (12) complications (bleeding, perforation, obstruction) required emergency surgery; (13) Pulmonary function tests FEV1 <50% of predicted value.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1056 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | three years

CONTACTS AND LOCATIONS:
Overall Officials: Guobin Wang, MD,PhD, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Kaixiong Tao, MD,PhD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China